CLINICAL TRIAL: NCT05021744
Title: Do Hand Grip Strength and Dexterity Predict of Respiratory Function in Neuromuscular Disease ?
Brief Title: Do Handgrip Strength and Dexterity Predict of Respiratory Function ?
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Collaborators: Medipol University (Other)
Responsible Party: Sponsor
Other Study IDs: BezmialemVU270717
Record Dates: First submitted 2021-08-04; First posted 2021-08-25 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Neuromuscular Diseases
MeSH Terms: conditions — Neuromuscular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Dysfunction due to weakness in respiratory muscles is one of the biggest problem that causes mortality and morbidity in neuromuscular diseases.Since the NMD have a crucial life-threading natural progression, many clinicians and researchers are trying to working out to increase life span and/or quality of life with medical and rehabilitative approaches.The relationship between upper extremity functions and respiratory functions in pediatric neuromuscular patients is still not clear. The clinician working with children with neuromuscular disease should be aware of the effects of muscle weakness and cognitive dysfunction on the respiratory system. Symptoms can be insidious and cause progressive loss of function, respiratory failure, and even death

DETAILED DESCRIPTION:
Background:Neuromuscular diseases are acquired or hereditary diseases that affect the function of the muscles in our body caused by the nerves not sending information to your muscles and/or problems with the muscles not working properly.

Objective:The aim of our study is to discover more cost-effective and practical tools to predict respiratory function losses that may be a significant problem in children with neuromuscular disease.

Methods: Hand grip strength and dexterity of children with neuromuscular disease were measured using the dynamometer and the nine-hole-peg-test respectively. The Vignos and Brooke Upper Extremity Functional Scales were used to evaluate functional status for patient recruitment.Respiratory function parameters:forced vital capacity (FVC), forced expiratory volume in one second (FEV1) and peak expiratory flow(PEF) were evaluated with spirometry.

ELIGIBILITY:
Inclusion Criteria:

* to be diagnosed with NMD
* to be in Stage 5 or below according to the Vignos scale (walking without assistance)
* to be between Stage 1-4 according to the Brooke scale.

Exclusion Criteria:

* Patients with severe systemic disease, ambulatory problem, cognitive problem, and upper extremity deformity were excluded

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Our study was carried out with 30 patients between the ages of 6-18 who were followed up with a diagnosis of neuromuscular disease.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2014-12-13 (Actual); Primary Completion 2015-12-13 (Actual); Study Completion 2016-01-01 (Actual)

PRIMARY OUTCOMES:
Respiratory Function Test | 1 day
  Respiratory function tests are noninvasive tests that show how well the lungs are working. The tests measure lung volume, capacity, rates of flow, and gas exchange.RFT measurements were made with the patients in the sitting position, with the nostrils closed with the help of a soft-headed clip that would not cause discomfort. The patients were asked to inhale and then exhale with the help of a cap attached to the spirometer device, which was placed in the mouth and ensured that there was no air leakage. Measurements were carried out in accordance with the standardization criteria determined jointly by the American Thoracic Society (ATS) and the European Respiratory Society (ERS). Cosmed Pony FX brand respiratory function test device was used.The percentages of the predicted values (percent) for forced expiratory volume in one second (FEV1), forced vital capacity (FVC), FEV1/FVC and peak expiratory flow (PEF) were used for statistical analysis.
Hand Grip Strength Test | 1 day
  Jamar hand dynamometer, which was recommended by the American Society of Hand Therapists and which has high validity and reliability in many studies and therefore accepted as the gold standard, was used in the measurement of hand grip strength of children. Participants were instructed to sit in a straight-backed chair with feet placed flat on the floor, shoulder abduction and neutral rotation, elbow flexion at 90 °, forearm and wrist in neutral position. Participants were asked to make an isometric contraction by squeezing the dynamometer with as much force as possible, making sure that only one contraction is made for each measurement. In all measurements, the score is evaluated in kilograms.
Hand Dexterity Assessment | 1 day
  Nine hole peg test was used to measure hand dexterity. Patients were asked to take nine wooden stick, one by one, from container, place them into holes, then collect them from the holes and put them back in the container. The board should be positioned in the patient's midline. The hand that is not evaluated should hold the edge of the board and provide stability. Times to complete the test are recorded with stopwatch in seconds

SECONDARY OUTCOMES:
Brooke Upper Extremity Functional Scale | 1 day
  The Brooke Upper Extremity Scale is a 6-point scale that allows classification of upper extremity function and also helps document progression.
  Functional Grades: Arms and Shoulders:
  Standing with arms at the sides, the patient can abduct the arms in a full circle until they touch above the head.
  The patient can raise the arms above the head only by flexing the elbow or by using accessory muscles (i.e. by shortening the circumference of the movement) The patient cannot raise hands above the head, but can raise an 8-oz. glass of water to the mouth (using both hands if necessary).
  The patient can raise hands to mouth, but cannot raise 8 oz. glass of water to the mouth The patient cannot raise hands to the mouth, but can use the hands to hold a pen or to pick up pennies from a table.
  The patient cannot raise hands to the mouth and has no useful function of the hands.
Vignos Functional Scale | 1 day
  In order to determine the patients to be included in the study, the ambulation levels of the patients were evaluated with the Vignos scale.
  Vignos scale for lower extremities
  1. Walks and climbs stairs without assistance
  2. Walks and climbs stair with aid of railing
  3. Walks and climbs stairs slowly with aid of railing (over 25 seconds for 8 standard steps)
  4. Walks unassisted and rises from chair but cannot climb stairs
  5. Walks unassisted but cannot rise from chair or climb stairs
  6. Walks only with assistance or walks independently with long leg braces
  7. Walks in long leg braces but requires assistance for balance
  8. Stands in long leg braces but unable to walk even with assistance
  9. Is in a wheelchair
  10. Is confined to a bed

CONTACTS AND LOCATIONS:
Overall Officials: Aysel Yıldız Ozer, Dr., Study Chair — Marmara University

IPD SHARING:
Plan to Share IPD: No